CLINICAL TRIAL: NCT01739179
Title: Laparoscopically Assisted Ventriculoperitoneal Shunt Placement: A Prospective, Randomized Two-arm Study
Brief Title: Keyhole Surgery for the Positioning of the Distal Catheter in Ventricular Peritoneal Shunt Placement
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 199/06
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Ventricular Peritoneal Shunt; Shunt Complications; Shunt Failure; Randomized Controlled Trial
Keywords: Ventricular peritoneal Shunt; Shunt Complications; Shunt Failure; Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: VP Shunt Surgery for laparoscopic insertion of the peritoneal catheter
  Interventions: Procedure: VP Shunt Surgery for laparoscopic insertion of the peritoneal catheter
- 2: VP Shunt Surgery for open insertion of the peritoneal catheter
  Interventions: Procedure: VP Shunt Surgery for open insertion of the peritoneal catheter

INTERVENTIONS:
Procedure: VP Shunt Surgery for laparoscopic insertion of the peritoneal catheter — Patients in this Study Arm will receive a VP Shunt inserted laparoscopically
  Groups: 1
Procedure: VP Shunt Surgery for open insertion of the peritoneal catheter — Patients in this Study Arm will receive a VP Shunt inserted openly
  Groups: 2

SUMMARY:
Ventriculoperitoneal shunting (VPS) was first described at the beginning of the 20th century as a diversionary procedure in patients with a hydrocephalus. After the introduction of silastic catheters in the 1970's this method became the treatment of choice for children and adults with communicating hydrocephalus. The average patient necessitating VPS will undergo at least two shunt revisions every three years, with some patients requiring more than twenty revisions within the first year. Therefore, any technical improvement with a positive impact on the revision rate not only benefits the patient through a reduction of the surgical burden but may also have economic advantages.

Distal shunt failures - either due to improper placement or secondary dislocation of the distal catheter out of the peritoneal cavity - have been reported in 10-30% of cases. Catheter placement in obese patients and in patients with adhesions owing to previous abdominal surgery remains challenging. Most neurosurgeons will carry out a mini-laparotomy to allow for the placement of the distal catheter end within the peritoneal cavity, which rarely requires the help of a general or visceral surgeon.

An alternative to laparotomy is the laparoscopic placement of the peritoneal catheter in VPS. Retrospective series have since shown the safety of this procedure and suggested an advantage of laparoscopic VPS in terms of operation duration, length of hospital stay and the rate of distal (and thus potentially overall) shunt dysfunction.

The evidence concerning the effect of laparoscopic surgery for VPS placement is so far based on non-randomized studies, in which a selection bias may have influenced the outcomes.

DETAILED DESCRIPTION:
Background

Ventriculoperitoneal shunting (VPS) as diversionary procedure in patients with hydrocephalus was first described in 1908. After the introduction of silastic catheters during the 1970s this method has become the treatment of choice for children and adults with communicating hydrocephalus. However, the average patient having had VPS will undergo 2.1 shunt revisions every 3 years of life, with a wide range from no revisions during the first decade to up to 21 revisions within the first year. For this reason technical improvements impacting positively on the revision rate and on the surgical burden are strongly needed.

In the standard VPS procedure the proximal part of the shunt is first placed in one of the lateral ventricles. The distal part of the shunt is then tunneled subcutaneously from the head to the abdomen, where 20-25 cm of the distal catheter and the tip are introduced in the peritoneal cavity through a paraumbilical mini-laparotomy. The intraperitoneal placement of the distal catheter is performed blindly, whereby the tip of the catheter is directed caudally in direction of the pelvis in order to avoid kinking and potential strangulation of the catheter. In this setting the functionality of the system can be estimated by feeling the resistance to out- and inflow while manually pumping the reservoir near the valve at the cranial level.

Distal shunt failure has been reported to occur in 10-30% of cases. Secondary dislocation of the peritoneal catheter in the subcutaneous tissue or its improper placement in the peritoneal cavity during the procedure both contribute to this high shunt failure rate. Furthermore, blind catheter placement in obese patients and in patients with adhesions from previous abdominal surgery can be a challenge and may lead to injuries of the intra-abdominal organs.

In 1993, Bassauri et al reported on the laparoscopic placement of the peritoneal catheter in VPS. Since then several, small retrospective series have shown good results in laparoscopic VPS, both in terms of efficacy and safety, in adults and in children. Two larger series were published recently. Schubert et al. reported a prospective study on 50 adult patients using the laparoscopically assisted peritoneal shunt insertion. A retrospective cohort of 50 matched patients served as a control. They reported no intraoperative complications, a longer operation time in the laparoscopic group (59 versus 49 minutes), 2 malfunctions (4%) and 1 infection in the laparoscopic group (2%) and 6 malfunctions (12%) and 6 infections (12%) in the historic cohort, the difference being statistically significant in favour of the laparoscopic group. In the most recent and largest series published to date, Bani et al. report on their experience with 151 patients, where the peritoneal catheter was implanted using a laparoscopic technique. They also used a retrospective cohort of 50 non-laparoscopy patients as a control. The operation time was slightly longer using the laparoscopic technique (35-130 versus 30-120 minutes), the infection rate was 2% in both groups. They describe no dislocation of the distal catheter in the abdominal wall and no malpositioning of the distal catheter in the laparoscopic group and 4 such cases in the non-laparoscopy group (8%).

In summary, these non-randomized trials suggest the safety of the procedure. The laparoscopic technique offers at least theoretically some significant advantages over the standard technique. The laparoscopic introduction of the peritoneal catheter allows for intra-abdominal inspection, lyses of adhesions whenever necessary, confirmation of the catheter position, and the visual assessment of cerebrospinal fluid (CSF) flow through the catheter tip during the procedure. Due to the minimal trauma to the abdominal wall the laparoscopic access also has the potential of reducing postoperative adhesions, wound complications and the overall postoperative morbidity. Despite these theoretical advantages, however, comparative, randomized data are lacking and ventriculoperitoneal shunting is still performed through a minilaparotomy in the vast majority of neurosurgical centres. The absence of scientific evidence favouring the laparoscopic technique, the lack of training of neurosurgeons in laparoscopic techniques and the potential prolongation of the operating time (and potentially a higher risk of infection) are probably the main reasons to explain why the shift to the laparoscopic technique has not yet taken place. Also, theoretically, the inflation of the peritoneal cavity for laparoscopy could potentially generate an acute hydrocephalus (e.g. during a distal revision) due to the elimination of the pressure gradient necessary to obtain flow of CSF into the peritoneal cavity.

These potential limitations warrant, in our view, a prospective, randomized, controlled trial comparing the standard (minilaparotomy) technique. The demonstration of the superiority of the laparoscopic technique in a prospective, randomized study has the potential of changing the standard of care for patients with hydrocephalus needing shunting.

Methods

120 patients scheduled for VPS surgery were randomised for laparoscopic or open insertion of the peritoneal catheter. The primary endpoint was the rate of overall shunt complication/failure after 12 months. Secondary endpoints were distal shunt failure rate at 6 weeks, 6 months and 12 months, overall complication/failure at 6 weeks and 6 months, duration of surgery and hospitalisation, and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* newly diagnosed hydrocephalus needing VP Shunt according to a board certified neurosurgeon
* Patients with shunt-malfunction needing VP Shunt revision and replacement of the peritoneal catheter
* Written Informed Consent

Exclusion Criteria

* Age younger than 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomized are all patients who are 18 years or older; who are treated at the Department of Neurosurgery, Inselspital Bern; who are diagnosed with a Hydrocephalus and need a VP Shunt; Patients who have a Shunt malfunction and Patient who have given the written approval (informed consent)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with overall shunt failure | 12 months

SECONDARY OUTCOMES:
Number of patients with distal shunt failure | 6 Weeks, 6 Months, 12 Months
Number of days to resumption of full oral food intake | 7 Days
Amount of analgesic (NSAID) drug intake as evaluated on day 5 postoperatively, measured in mg | 5 Days
Duration of Operation | 10 hours
Duration of Hospital Stay | 20 Days
Time to recover full mobility | 15 Days
Number of patients with correct proximal and distal catheter positioning | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe E Schucht, MD, Principal Investigator — Department of Neurosurgery
Locations (1):
- Department of Neurosurgery, Bern, Switzerland

REFERENCES:
- [Result] Raimondi AJ, Matsumoto S. A simplified technique for performing the ventriculo-peritoneal shunt. Technical note. J Neurosurg. 1967 Mar;26(3):357-60. doi: 10.3171/jns.1967.26.3.0357. No abstract available. PMID 6019744
- [Result] Ames RH. Ventriculo-peritoneal shunts in the management of hydrocephalus. J Neurosurg. 1967 Dec;27(6):525-9. doi: 10.3171/jns.1967.27.6.0525. No abstract available. PMID 6065126
- [Result] Grosfeld JL, Cooney DR, Smith J, Campbell RL. Intra-abdominal complications following ventriculoperitoneal shunt procedures. Pediatrics. 1974 Dec;54(6):791-6. No abstract available. PMID 4431676
- [Result] Khosrovi H, Kaufman HH, Hrabovsky E, Bloomfield SM, Prabhu V, el-Kadi HA. Laparoscopic-assisted distal ventriculoperitoneal shunt placement. Surg Neurol. 1998 Feb;49(2):127-34; discussion 134-5. doi: 10.1016/s0090-3019(97)00357-1. PMID 9457261
- [Result] Abu-Dalu K, Pode D, Hadani M, Sahar A. Colonic complications of ventriculoperitoneal shunts. Neurosurgery. 1983 Aug;13(2):167-9. doi: 10.1227/00006123-198308000-00011. PMID 6888697
- [Result] Wilson CB, Bertan V. Perforation of the bowel complicating peritoneal shunt for hydrocephalus. Report of two cases. Am Surg. 1966 Sep;32(9):601-3. No abstract available. PMID 5916956
- [Result] Basauri L, Selman JM, Lizana C. Peritoneal catheter insertion using laparoscopic guidance. Pediatr Neurosurg. 1993 Mar-Apr;19(2):109-10. doi: 10.1159/000120711. PMID 8443096
- [Result] Cuatico W, Vannix D. Laparoscopically guided peritoneal insertion in ventriculoperitoneal shunts. J Laparoendosc Surg. 1995 Oct;5(5):309-11. doi: 10.1089/lps.1995.5.309. PMID 8845504
- [Result] Bani A, Hassler WE. Laparoscopy-guided insertion of peritoneal catheters in ventriculoperitoneal shunt procedures: analysis of 39 children. Pediatr Neurosurg. 2006;42(3):156-8. doi: 10.1159/000091858. PMID 16636616
- [Result] Schievink WI, Wharen RE Jr, Reimer R, Pettit PD, Seiler JC, Shine TS. Laparoscopic placement of ventriculoperitoneal shunts: preliminary report. Mayo Clin Proc. 1993 Nov;68(11):1064-6. doi: 10.1016/s0025-6196(12)60899-4. PMID 8231270
- [Result] Reardon PR, Scarborough TK, Matthews BD, Marti JL, Preciado A. Laparoscopically assisted ventriculoperitoneal shunt placement using 2-mm instrumentation. Surg Endosc. 2000 Jun;14(6):585-6. doi: 10.1007/s004640020078. PMID 10890971
- [Result] Kirshtein B, Benifla M, Roy-Shapira A, Merkin V, Melamed I, Cohen Z, Cohen A. Laparoscopically guided distal ventriculoperitoneal shunt placement. Surg Laparosc Endosc Percutan Tech. 2004 Oct;14(5):276-8. doi: 10.1097/00129689-200410000-00009. PMID 15492657
- [Derived] Schucht P, Banz V, Trochsler M, Iff S, Krahenbuhl AK, Reinert M, Beck J, Raabe A, Candinas D, Kuhlen D, Mariani L. Laparoscopically assisted ventriculoperitoneal shunt placement: a prospective randomized controlled trial. J Neurosurg. 2015 May;122(5):1058-67. doi: 10.3171/2014.9.JNS132791. Epub 2014 Dec 23. PMID 25534231